CLINICAL TRIAL: NCT05330013
Title: Pilot Study to Evaluate the Effect of Inflammation in Heart Failure
Brief Title: The Effect of Inflammation in Heart Failure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left NIH
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10000710; 000710-H
Record Dates: First submitted 2022-04-14; First posted 2022-04-15 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Myocardial Dysfunction; Heart Failure; Inflammation
Keywords: Dapagliflozin; Hfpef; Cardiac MRI; NLRP3 Inflammasome; Perfusion
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — dapagliflozin; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Healthy volunteers who are age and sex matched
  Interventions: Device: MRI scan; Device: CMR imaging
- Subjects with HFpEF (Experimental): Subjects are defined as patients with a diagnosis of HFpEF clinically confirmed by a licensed physician or advanced practitioner who meet the inclusion and exclusion criteria and are able to provide informed consent.
  Interventions: Drug: Dapagliflozin; Device: MRI scan; Device: CMR imaging

INTERVENTIONS:
Drug: Dapagliflozin — Subjects will be instructed to take dapagliflozin 10 mg once daily for 6 months (with or without food).
  Arms: Subjects with HFpEF
Device: MRI scan — For subjects, depending on the subject's heart rate, base, mild, or apex short-axis slices will be acquired during the first pass of the contract (60 measurements).
Device: CMR imaging — Enrolled subjects will undergo stress vasodilator and rest perfusion CMR

SUMMARY:
Background:

Heart failure is a serious health condition. Researchers believe inflammation plays a role. They want to see if adding an additional heart drug to a person s treatment can help treat heart failure with preserved ejection fraction (HFpEF).

Objective:

To learn if chronic inflammation is high in heart failure and if taking dapagliflozin along with the standard of care medicines for 6 months will reduce inflammation and improve heart function in people with HFpEF.

Eligibility:

People aged 18 and older who have heart failure and qualify for dapagliflozin therapy. Healthy adult volunteers are also needed.

Design:

* Participants will be screened with:

  * Medical history
  * Physical exam
  * Heart function tests
  * X-ray scans of the heart and blood vessels. They may receive medicines to slow their heart rate or make their heart blood vessels bigger. An intravenous (IV) catheter will be placed in their arm to inject contrast.
  * Blood and urine tests
* Participants will have up to 3 study visits. Some screening tests will be repeated.

Participants will take one tablet of the study drug daily for 6 months.

-Participants will have an imaging scan of their heart and blood vessels. They will receive a contrast and stress medicine through an IV to view blood supply.

Participants will have a stress test that measures exercise ability. They will wear sticky pads on their chest, a blood pressure cuff, and a mask. They will also have a 6-Minute Walk Test.

Participants will complete questionnaires about their symptoms and their health.

Participants may be on the study for up to 6 months. They will have a follow-up phone call 1 month after treatment ends.

...

DETAILED DESCRIPTION:
Study Description:

Heart failure (HF) remains a significant public health burden. Unlike heart failure with reduced ejection fraction (HFrEF), heart failure with preserved ejection fraction (HFpEF) currently does not have any effective therapies, suggesting incomplete understanding of the underlying mechanisms of the syndrome. Chronic inflammation has been postulated to be one of the central mechanisms in HFpEF pathogenesis. In this pilot study to be conducted at the NIH Clinical Center, we propose to examine the role of the NLRP3 inflammasome- IL-1 pathway in HFpEF and evaluate whether treatment using the sodium glucose co-transport 2 (SGLT2) inhibitor dapagliflozin can attenuate NLRP3 inflammasome activation.

Objectives:

* To test the hypothesis that macrophage NLRP3 inflammasomeactivation is upregulated in subjects with HFpEF compared to healthy controls and that NLRP3 inflammasome activation will be attenuated by dapagliflozin therapy
* To test the hypothesis that pro-inflammatory signatures in peripheral blood mononuclear cells (PBMCs) will be increased in HFpEF compared to healthy controls and that they will be attenuated by dapagliflozin therapy
* To test the hypothesis that macrophage NLRP3 inflammasome activation associates with perturbances in myocardial perfusion, structure, and function and that attenuation of NLRP3 inflammasome activation with dapagliflozin therapy will associate with improvement in myocardial perfusion, myocardial structure, and function
* To test the hypothesis that NLRP3 inflammasome activation is inversely associated with maximum oxygen consumption (VO2max), exercise functional status, and symptoms in HFpEF and that attenuation of NLRP3 inflammasome activation with dapagliflozin therapy will associate with improvement in VO2max, exercise functional status, and symptoms.

Endpoints:

Primary outcome will be:

-IL-1 beta, a measure of NLRP3 inflammasome activation, from macrophages in subjects with HFpEF compared to healthy controls.

Secondary outcomes will be:

* Delineation of the differences in PBMC gene expression profiles measured by RNA sequencing and in immunophenotyping signatures measured by flow cytometry in subjects with HFpEF compared to healthy controls. The effect of dapagliflozin on these immunological profiles will also be determined in the HFpEF study subjects.
* Myocardial perfusion (on CMR), left ventricular mass (on CMR), diastolic function (on echocardiogram), myocardial mechanics (on echocardiogram and CMR), myocardial edema and inflammation, and interstitial fibrosis (on CMR) in subjects with HFpEF compared to healthy controls and in response to dapagliflozin therapy.

Exploratory outcomes will be:

- VO2max, symptoms and exercise functional status in HFpEF compared to healthy controls and in response to dapagliflozin therapy.

ELIGIBILITY:
* INCLUSION CRITERIA

Subjects of both genders will be considered for inclusion in this study. There will be no racial, ethnic, or gender discrimination.

Affected Subjects:

* 18years of age or older
* Diagnosed with HFpEF clinically confirmed by licensed physician or advanced practitioner
* Signs and symptoms of HFpEF
* LVEF >= 50% on echocardiography from screening visit
* Left ventricular hypertrophy (interventricular septal thickness (Bullet) 1cm) or enlarged left atrial volume ( (Bullet)34ml/m2) on echocardiography from screening visit
* NT-proBNP > 300pg/mL

Healthy Controls:

Females and males 18 years of age or older

EXCLUSION CRITERIA:

Affected Subjects:

* Pregnant or lactating women
* Acute coronary syndrome, cardiac surgery or percutaneous coronary intervention within past 6 months
* Atrial fibrillation
* Coronary artery disease with >= 50% stenosis in the left main, left anterior descending artery, left circumflex artery, or right coronary artery on CCTA from screening visit
* Infiltrative cardiomyopathy by diagnosis or imaging

  -> Moderate valvular stenosis on screening echocardiography
* Diagnosis of an inflammatory disease (including psoriasis, psoriatic arthritis, rheumatoid arthritis, lupus, inflammatory bowel disease, HIV)
* Currently taking an SGLT2 inhibitor
* Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73m^2 body surface area according to the Modification of Diet in Renal Disease criteria
* Subjects with a contraindication to MRI scanning will not receive the CMR assessment.

These contraindications include subjects with the following devices:

i. Central nervous system aneurysm clips

ii. Implanted neural stimulator

iii. Implanted cardiac pacemaker or defibrillator

iv. Cochlear implant

v. Ocular foreign body (e.g. metal shavings)

vi. Implanted Insulin pump

vii. Metal shrapnel or bullet

* History of seizures or taking anti-epileptic medications
* History of serious hypersensitivity to dapagliflozin
* History of diabetic ketoacidosis
* Inability to provide informed consent

Healthy Controls:

* History of HF
* Acute coronary syndrome, cardiac surgery or percutaneous coronary intervention within past 6 months
* Coronary artery disease with >= 50% stenosis in the left main, left anterior descending artery, left circumflex artery, or right coronary artery on CCTA
* Diagnosis of an inflammatory disease (including psoriasis, psoriatic arthritis, rheumatoid arthritis, lupus, inflammatory bowel disease, HIV)
* Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73m^2 body surface area according to the Modification of Diet in Renal Disease criteria
* Pregnant women and lactating women
* Subjects with a contraindication to MRI scanning will not receive the CMR assessment.

These contraindications include subjects with the following devices:

viii. Central nervous system aneurysm clips

ix. Implanted neural stimulator

x. Implanted cardiac pacemaker or defibrillator

xi. Cochlear implant

xii. Ocular foreign body (e.g. metal shavings)

xiii. Implanted Insulin pump

xiv. Metal shrapnel or bullet

* History of seizures or taking anti-epileptic medications
* Inability to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
IL-1 beta levels | 6 months
  IL-1 beta, a measure of NLRP3 inflammasome activation, from macrophages in subjects with HFpEF compared to healthy controls

SECONDARY OUTCOMES:
Change in CMR, ECHO in affected vs healthy individuals | 2.5 years
  1. Myocardial perfusion(CMR), 2. Left ventricular mass(CMR), 3. Diastolic function (ECHO), 4. Myocardial mechanics (ECHO, CMR), 5. Myocardial edema and inflammation, and interstitial fibrosis(CMR) Compared to both group and in response to dapagliflozin therapy
Immunological profiles in affected vs healthy individuals | 2.5 years
  Delineation of the differences in PBMC gene expression profiles measured by RNA sequencing and in immunophenotyping signatures measured by flow cytometry in subjects with HFpEF compared to healthy controls. The effect of dapagliflozin on these immunological profiles will also be determined in the HFpEF study subjects

CONTACTS AND LOCATIONS:
Overall Officials: Wunan Y Zhou, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kim SR, Lee SG, Kim SH, Kim JH, Choi E, Cho W, Rim JH, Hwang I, Lee CJ, Lee M, Oh CM, Jeon JY, Gee HY, Kim JH, Lee BW, Kang ES, Cha BS, Lee MS, Yu JW, Cho JW, Kim JS, Lee YH. SGLT2 inhibition modulates NLRP3 inflammasome activity via ketones and insulin in diabetes with cardiovascular disease. Nat Commun. 2020 May 1;11(1):2127. doi: 10.1038/s41467-020-15983-6. PMID 32358544
- [Background] Brown AJM, Gandy S, McCrimmon R, Houston JG, Struthers AD, Lang CC. A randomized controlled trial of dapagliflozin on left ventricular hypertrophy in people with type two diabetes: the DAPA-LVH trial. Eur Heart J. 2020 Sep 21;41(36):3421-3432. doi: 10.1093/eurheartj/ehaa419. PMID 32578850
- [Background] Anker SD, Butler J, Filippatos G, Ferreira JP, Bocchi E, Bohm M, Brunner-La Rocca HP, Choi DJ, Chopra V, Chuquiure-Valenzuela E, Giannetti N, Gomez-Mesa JE, Janssens S, Januzzi JL, Gonzalez-Juanatey JR, Merkely B, Nicholls SJ, Perrone SV, Pina IL, Ponikowski P, Senni M, Sim D, Spinar J, Squire I, Taddei S, Tsutsui H, Verma S, Vinereanu D, Zhang J, Carson P, Lam CSP, Marx N, Zeller C, Sattar N, Jamal W, Schnaidt S, Schnee JM, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Preserved Trial Investigators. Empagliflozin in Heart Failure with a Preserved Ejection Fraction. N Engl J Med. 2021 Oct 14;385(16):1451-1461. doi: 10.1056/NEJMoa2107038. Epub 2021 Aug 27. PMID 34449189
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000710-H.html